CLINICAL TRIAL: NCT06130306
Title: Electrical Pudendal Nerve Stimulation Versus Pelvic Floor Muscle Training Plus Transanal Electrical Stimulation for Post-Radical Prostatectomy Incontinence: A Propensity Score Matching Analysis
Brief Title: A PSM Analysis to Evaluate Electrical Pudendal Nerve Stimulation for PPI
Status: Completed | Type: Observational
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Shanghai Pudong Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: PWRq2022-47
Record Dates: First submitted 2023-11-05; First posted 2023-11-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2023-08

CONDITIONS: Urinary Incontinence Following Surgical Procedure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electrical Pudendal Nerve Stimulation Group: Electrical Pudendal Nerve Stimulation
  Interventions: Procedure: electrical pudendal nerve stimulation
- Pelvic Floor Muscle Training Group: Pelvic Floor Muscle Training Plus Transanal Electrical Stimulation
  Interventions: Procedure: pelvic floor muscle training combined with transanal electrical stimulation

INTERVENTIONS:
Procedure: electrical pudendal nerve stimulation — The patient was positioned prone post-micturition. Long needles (0.40 Х 100 mm) were inserted perpendicularly, 1 cm bilateral to the sacrococcygeal joint, to a depth of 80-90 mm, eliciting sensations referred to the urethra or anus. The lower points, 1 cm bilateral to the coccyx tip, received oblique insertion of longer needles (0.40 Х 125 mm) toward the ischiorectal fossa (90-110 mm depth), inducing sensations precisely to the urethra. Connected to a G6805-2 Multi-Purpose Health Device, the ipsilateral needles created an electric loop, with the upper as anode and lower as cathode. Direct electrical stimulation (2.5 Hz, 25~35 mA) for 45 minutes targeted the pudendal nerve, thrice weekly for a minimum of 8 weeks. The treatment plan remains ongoing until the patient opts to discontinue voluntarily.
  Groups: Electrical Pudendal Nerve Stimulation Group
Procedure: pelvic floor muscle training combined with transanal electrical stimulation — Electromyogram BF-assisted PFMT (using a nerve function reconstruction treatment system [AM1000B; Shenzhen Creative Industry Co. Ltd, China]) and following TES (using a neuromuscular stimulation therapy system (PHENIX USB 4, Electronic Concept Lignon Innovation, France)) at a current intensity of < 60 mA (as high as possible to get a PFM contraction) and frequencies of 15 Hz and 85 Hz (alternate 3-minute periods of stimulation) were performed by a specially trained therapist, 20 minutes each time, respectively (a total of 40 minutes), 3 times a week for a total of 8 weeks. The patients also conducted 30 maximal high-intensity PFM contractions for 2-6 seconds (with 2-6 seconds rest), 3 sessions every day at home for a total of 8 weeks. If the patient is willing, the treatment plan can continue until the patient voluntarily decides to stop.
  Groups: Pelvic Floor Muscle Training Group

SUMMARY:
The goal of this propensity score matching study is to compare the posttreatment outcomes of post-radical prostatectomy Incontinence patients undergoing either electrical pudendal nerve stimulation or pelvic floor muscle training combined with transanal electrical stimulation.

DETAILED DESCRIPTION:
Prostate cancer is the predominant form of cancer in older males. Radical prostatectomy (RP) is the sole treatment that enhances both overall survival and cancer-specific survival.Urinary incontinence remains a major morbidity associated with this procedure, greatly affecting patient satisfaction following RP. Extant research underscores the efficacy of pelvic floor muscle training (PFMT) in improving the strength and function of specific pelvic floor muscles, causing hypertrophy of peri-urethral striated muscles, thereby increasing the external mechanical pressure on the urethra. Another promising physiotherapy for post-radical prostatectomy incontinence (PPI) is electrical pudendal nerve stimulation (EPNS). An increasing body of research focuses on comparing continence restoration outcomes between PFMT and various electrical stimulations. However, such studies encompass cases with multiple pathological characteristics, and the reported data might not be considered representative or applicable to other populations due to overlooked confounding factors or selection bias. Thus, the investigators intend to conduct a propensity score matching (PSM) study aiming to compare the posttreatment outcomes of patients undergoing either EPNS or PFMT combined with TES, while ensuring a well-balanced control for confounding factor.

ELIGIBILITY:
Inclusion Criteria:

* Onset of urinary incontinence at least 1 month post-RP
* Minimum two documented incontinence episodes per week in a 7-day bladder diary
* Pathological confirmation of no residual cancer post-RP

Exclusion Criteria:

* High pathological risk factors (e.g., lymph node metastasis, resection margin involvement, bulky tumors)
* Preoperative incontinence
* Prior anticholinergic treatment
* Urinary tract infection or hematuria
* Postvoid residual volume exceeding 100 ml (determined by bladder ultrasound)
* Neurological disorders
* Urethral stricture

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18-80 with post-radical prostatectomy incontinence treated at 3 tertiary academic medical centers between 2012 and 2020 were retrieved.
Sampling Method: Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire-short form score (ICIQ-SF) | T0 (baseline); T1 (day after 24th treatment); T2 (day after 36th treatment); T3 (day after 48th treatment); T4 (day after 60th treatment); T5 (day after 72nd treatment).
  The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) is a validated and widely used questionnaire to assess and measure the impact of urinary incontinence on an individual's quality of life. This part includes a set of simple questions related to urinary incontinence symptoms, which the individual answers. The questions address the type and frequency of incontinence episodes, as well as their impact on daily life. The higher the score, the more severe the condition.

SECONDARY OUTCOMES:
Pad-counting Score | T0 (baseline); T1 (day after 24th treatment); T2 (day after 36th treatment); T3 (day after 48th treatment); T4 (day after 60th treatment); T5 (day after 72nd treatment).
  the number of urine pad consumption in 24 hours.The higher the score, the more severe the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Siyou Wang, Principal Investigator — Shanghai research institute of acupuncture and meridian
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
If necessary, contact Dr. Siyou Wang to provide the original data.

REFERENCES:
- [Derived] Li T, Wang S, Chen Q, Lv T, Huang Z. Electrical pudendal nerve stimulation versus pelvic floor muscle training with transrectal electrical stimulation for post-radical prostatectomy incontinence: a cohort study. Sci Rep. 2025 Nov 24;15(1):41603. doi: 10.1038/s41598-025-25567-3. PMID 41286037